CLINICAL TRIAL: NCT01715792
Title: Risk of Solid Organ Transplant Rejection Following Vaccination With Pandemrix™ in the United Kingdom
Brief Title: Assess the Risk of Solid Organ Transplant Rejection Following Vaccination With Pandemrix™ in UK
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116602
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Influenza
Keywords: Solid organ transplant rejection; United Kingdom; Influenza; H1N1; Pandemrix™
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Group 1: Subject defined as acceptable in the CPRD GOLD with at least one solid organ transplant rejection reported during the overall study period (01 September to 31 October 2010).
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data extraction from the CPRD GOLD and HES, and additional data obtained from complementary information provided by the GPs using a standardised questionnaire.

SUMMARY:
This study aims to assess the risk of solid organ transplant (SOT) rejection following vaccination with Pandemrix™ and/ or seasonal influenza vaccination.

DETAILED DESCRIPTION:
Data on the safety of pandemic H1N1 vaccination in transplanted patients is relatively limited; to date, although some studies showed transient increases in alloreactivity, there is no evidence that H1N1 vaccines caused clinical rejection or organ dysfunction. In addition, studies have shown that influenza infection is a known independent risk factors for rejection. Considering that transplant recipients are a target population for immunisation with future pandemic vaccines, it is important to investigate the risk of rejection following vaccination in this patient population.

Using the self-controlled case series design that allows to control implicitly for potential confounding factors, this study aims at investigating the risk of solid organ transplant rejection (liver, kidney, lung, heart, pancreas) following vaccination with Pandemrix™ in the United Kingdom Clinical Practice Research Datalink GP Online Database (CPRD GOLD). Data from the Hospital Episodes Statistics database will also be used. The effect of seasonal influenza vaccination and of various infections including influenza H1N1 will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Subject defined as acceptable in the CPRD GOLD.
* Subject with at least one solid organ transplant rejection reported in the CPRD GOLD and/or HES during the overall study periods (01 September 2006 to 31 October 2010).

Exclusion Criteria:

• Subject from HES matched to more than one subject in the CPRD GOLD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subject defined as acceptable in the CPRD GOLD with at least one solid organ transplant rejection reported during the overall study periods (01 September 2006 to 31 October 2010).
Sampling Method: Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the risk of solid organ transplant rejection (liver, kidney, lung, heart, pancreas). | Within one month after vaccination with Pandemrix™ (from 01 October 2009 to 31 October 2010).
  Assessed by case data collection from CPRD GOLD and HES, and additional data obtained from complementary information provided by the GPs using a standardised questionnaire.

SECONDARY OUTCOMES:
Assessment of the risk of solid organ transplant rejection (liver, kidney, lung, heart, pancreas). | Within two months after vaccination with Pandemrix™ ( from 01 October 2009 to 31 October 2010).
  Assessed by case data collection from CPRD GOLD and HES, and additional data obtained from complementary information provided by the GPs using a standardised questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Cohet C, Haguinet F, Dos Santos G, Webb D, Logie J, Lc Ferreira G, Rosillon D, Shinde V. Effect of the adjuvanted (AS03) A/H1N1 2009 pandemic influenza vaccine on the risk of rejection in solid organ transplant recipients in England: a self-controlled case series. BMJ Open. 2016 Jan 28;6(1):e009264. doi: 10.1136/bmjopen-2015-009264. PMID 26823177